CLINICAL TRIAL: NCT01283984
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled AZD2115 After Single Ascending Doses in Healthy Male Subjects
Brief Title: AZD2115 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Carin Jorup / Medical Science Director, AstraZeneca R&D Lund
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3060C00001
Record Dates: First submitted 2011-01-05; First posted 2011-01-26 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Disease Causing Persistent Narrowing of the Airways
Keywords: Safety; tolerability; healthy; inhaled; respiratory disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): AZD2115
  Interventions: Drug: AZD2115
- 2 (Placebo Comparator): Placebo to AZD2115
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2115 — Single dose, oral inhalation (nebuliser solution)
  Arms: 1
Drug: Placebo — Single dose, oral inhalation (nebuliser solution)
  Arms: 2

SUMMARY:
AZD2115 Single Ascending Dose Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms with spermicide, from the day of dosing until 3 months after dosing with the investigational product.
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be able to inhale from a Spira nebuliser according to given instructions

Exclusion Criteria:

* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome
* Any clinically important abnormalities in heart rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following:

  * PR (PQ) interval prolongation >200 ms (first degree AV block)
  * Intermittent second or third degree AV block (based on screening or pre-dose ECG)
  * Incomplete, full or intermittent bundle branch block (QRS <110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy)
  * Abnormal T wave morphology, particularly in the protocol defined primary lead
  * Dropped beats
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD2115 and/or excipients
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Serum potassium concentration of <3.80 mmol/L on admission (Day -1)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the frequency of adverse events of inhaled single doses of AZD2115 | Measurements will be taken at screening
To evaluate the laboratory safety assessments of inhaled single doses of AZD2115 | Measurements will be taken at screening
To evaluate the vital signs of inhaled single doses of AZD2115 | Measurements will be taken at screening
To evaluate the physical examination of inhaled single doses of AZD2115 | Measurements will be taken at screening
To evaluate the ECG of inhaled single doses of AZD2115 | Measurements will be taken at screening
To evaluate the frequency of adverse events of inhaled single doses of AZD2115 | Measurements will be taken pre-dose
To evaluate the frequency of adverse events of inhaled single doses of AZD2115 | Measurements will be taken at multiple timelpoints during dosing day through to 48 hours post-dose
To evaluate the frequency of adverse events of inhaled single doses of AZD2115 | Measurements will be taken at follow up 7-13 days post dose.
To evaluate the laboratory safety assessments of inhaled single doses of AZD2115 | Measurements will be taken at pre-dose
To evaluate the laboratory safety assessments of inhaled single doses of AZD2115 | Measurements will be taken at multiple timelpoints during dosing day through to 48 hours post-dose
To evaluate the laboratory safety assessments of inhaled single doses of AZD2115 | Measurements will be taken at follow up 7-13 days post dose.
To evaluate the vital signs of inhaled single doses of AZD2115 | Measurements will be taken at pre-dose
To evaluate the vital signs of inhaled single doses of AZD2115 | Measurements will be taken at multiple timelpoints during dosing day through to 48 hours post-dose
To evaluate the vital signs of inhaled single doses of AZD2115 | Measurements will be taken at follow up 7-13 days post dose.
To evaluate the physical examination of inhaled single doses of AZD2115 | Measurements will be taken at pre-dose
To evaluate the physical examination of inhaled single doses of AZD2115 | Measurements will be taken at multiple timelpoints during dosing day through to 48 hours post-dose
To evaluate the physical examination of inhaled single doses of AZD2115 | Measurements will be taken at follow up 7-13 days post dose.
To evaluate the ECG of inhaled single doses of AZD2115 | Measurements will be taken at pre-dose
To evaluate the ECG of inhaled single doses of AZD2115 | Measurements will be taken at multiple timelpoints during dosing day through to 48 hours post-dose
To evaluate the ECG of inhaled single doses of AZD2115 | Measurements will be taken at follow up 7-13 days post dose.

SECONDARY OUTCOMES:
To assess the pharmacokinetics of a single dose of AZD2115 by assessment of area under the curve over the time (AUC) and maximum concentration (Cmax). | Frequent sampling occasions during study days, before and up to 48 h after dosing
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - FEV1 | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - potassium | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - glucose | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - systolic and diastolic blood pressure | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - pulse, heart rate | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.
To investigate the pharmacodynamic effects of inhaled single ascending doses of AZD2115 - QTcF | Measurements will be taken at screening, pre-dose and at multiple timelpoints during dosing day through to 48 hours post-dose and then again at follow up 7-13 days post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, UK, United Kingdom